CLINICAL TRIAL: NCT00589277
Title: Promoting Tobacco and Cancer Control: Message Framing for Telephone Quitline Callers
Brief Title: Message Framing for Telephone Quitline Callers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0705002661; R21CA127818 (NIH)
Record Dates: First submitted 2008-01-03; First posted 2008-01-09 (Estimated); Results first posted 2013-02-05 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Smoking; Nicotine Dependence
Keywords: Smoking; Tobacco; Message Framing
MeSH Terms: conditions — Smoking; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gain-Framed counseling & Gain-framed materials (Experimental): Novel messages for quitting smoking
  Interventions: Behavioral: Gain-Framed counseling & Gain-framed materials
- Standard care counseling + standard materials (Placebo Comparator): Standard care counseling + standard care print information
  Interventions: Behavioral: Standard care counseling + standard materials

INTERVENTIONS:
Behavioral: Gain-Framed counseling & Gain-framed materials — Novel messages for quitting smoking
  Arms: Gain-Framed counseling & Gain-framed materials
Behavioral: Standard care counseling + standard materials — Standard messages for quitting smoking
  Arms: Standard care counseling + standard materials

SUMMARY:
The purpose of this study is to compare gain-framed counseling + gain-framed materials" to standard care Quitline counseling + standard print materials. The investigators hypothesize that gain-framed counseling + gain-framed materials group will produce higher abstinence rates than standard care counseling and standard care information. The data in this study will be used to determine effect size estimates for a large scale study.

DETAILED DESCRIPTION:
This pilot study is meant to be translational (i.e., positive study results could easily translate to the actual practices of the NYS Smokers' Quitline) - as much as possible, the standard practices of the Quitline will be followed. In this context, a randomized pilot clinical trial comparing exclusively "Gain-framed counseling + gain-framed materials" to standard care Quitline counseling + standard print materials will be conducted with individuals calling the NYS Smokers' Quitline for assistance in quitting smoking. Following assessment of eligibility and informed consent, 2,500 smokers will be assisted by Specialists in either the YC or SC experimental conditions.

Consistent with the current practices of the Quitline, following the counseling intervention, participants will be mailed a package containing print materials encouraging smoking cessation, and participants eligible for Nicotine replacement therapy (NRT) will receive a 2-week supply of nicotine replacement medication. Consistent with Quitline practices, all callers will be required to set a "quit date" within 2 weeks of their initial call. A Quitline Specialist will initiate a follow-up call approximately 10 to 14 days after the print materials and NRT has been mailed. For callers receiving NRT, the manufacturer's suggested course of therapy (e.g., 8 weeks of NRT) will be recited to callers, and Quitline Specialists will suggest that callers use the money they save from not smoking to purchase additional NRT and/or that they check with their insurance carrier to see if additional NRT would be covered.

Participants will be assessed before receiving the gain-framed counseling + gain-framed materials or standard care counseling, immediately after receiving counseling, approximately 1 week after their quit date for those who receive NRT, and at a 3-month follow-up to see if the gain-framed counseling + gain-framed materials participants, as predicted, are more likely to promote smoking cessation. Several brief measures that assess potential mediator of treatment will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+ years)
* New York State residents
* English-speaking
* Current smokers who utilize Quitline services seeking quitting assistance for themselves

Exclusion Criteria:

* Callers who are enrolled in the Proactive Program for Medicaid/uninsured clients, or special programs through their insurance company or county

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2032 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin A Toll, Ph.D., Principal Investigator — Yale University
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] Toll BA, Martino S, Latimer A, Salovey P, O'Malley S, Carlin-Menter S, Hopkins J, Wu R, Celestino P, Cummings KM. Randomized trial: Quitline specialist training in gain-framed vs standard-care messages for smoking cessation. J Natl Cancer Inst. 2010 Jan 20;102(2):96-106. doi: 10.1093/jnci/djp468. Epub 2010 Jan 7. PMID 20056957

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care Counseling + Standard Care Print Information: Standard care counseling + standard care print information
- Gain-Framed Counseling: Callers were randomly assigned to receive gain-framed counseling messages and received newly developed, exclusively gain-framed NYSSQL printed materials by mail.
Period: Overall Study
Arm/Group | Standard Care Counseling + Standard Care Print Information | Gain-Framed Counseling
Started | 1222 | 810
Completed 2 Week Follow Up | 603 | 424
Completed 3 Month Follow Up | 762 | 524
Completed | 762 | 524
Not Completed | 460 | 286

BASELINE CHARACTERISTICS:
Groups:
- Standard Care Counseling: Standard care counseling + standard care print information
- Gain-Framed Counseling: Callers were randomly assigned to receive standard care counseling and materials or were exposed to gain-framed counseling statements and received newly developed, exclusively gain-framed NYSSQL printed materials by mail.
- Total: Total of all reporting groups
Arm/Group | Standard Care Counseling | Gain-Framed Counseling | Total
Number analyzed (Participants) | 1222 | 810 | 2032
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (13.9) | 47.2 (13.4) | 46.5 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 675 | 478 | 1153
  Male | 547 | 332 | 879

OUTCOME MEASURES:

1. Primary Outcome: Quit Attempt
Description: Percentage of those that self reported attempting to quit smoking at the 2 week follow up.
Time Frame: 2 week follow up
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Standard Care Counseling | Gain-Framed Counseling
Number analyzed (Participants) | 603 | 424
participants | 101 | 132

2. Secondary Outcome: 24 Hour Abstinence
Description: The number of survey respondents that had abstained from smoking at the 2 week follow up.
Time Frame: 2 week follow up
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Standard Care Counseling | Gain-Framed Counseling
Number analyzed (Participants) | 603 | 424
participants | 76 | 99

3. Secondary Outcome: 7 Day Abstinence
Description: The number of survey respondents that had abstained from smoking for 7 days at the 3 month follow up.
Time Frame: 3 month follow up
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Standard Care Counseling | Gain-Framed Counseling
Number analyzed (Participants) | 762 | 524
participants | 202 | 148

ADVERSE EVENTS:
Arm/Group | Standard Care Counseling | Gain-Framed Counseling
Serious Adverse Events (participants affected / at risk) | 0/1222 | 0/810
Other Adverse Events (participants affected / at risk) | 0/1222 | 0/810

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No